CLINICAL TRIAL: NCT00273442
Title: Assessing Cosopt Switch Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRN 05-007
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma; Exfoliation Syndrome; Glaucoma, Pigmentary
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Timolol; dorzolamide

INTERVENTIONS:
Drug: timolol maleate
Drug: dorzolamide/timolol maleate fixed combination

SUMMARY:
To assess the safety and efficacy of a cohort of patients switched to the dorzolamide/timolol maleate fixed combination because they are insufficiently controlled on latanoprost monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* adults with clinical diagnosis of POAG, pigment-dispersion or exfoliation glaucoma or ocular hypertension
* the IOP on latanoprost must be 31 mm Hg or less in both eyes, and 21 to 31 mm Hg inclusive in at least one eye at 08:00 AM
* visual acuity should be 20/200 or better in each eye

Exclusion Criteria:

* contraindications to study drugs
* anticipated change in systemic hypotensive therapy during the trial
* use of any corticosteroids by any route in the three months immediately prior to Visit 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Mark J. Weiss, MD, Principal Investigator; Douglas G. Day, MD, Principal Investigator — Omni Eye Services; Sriram Sonty, MD, FACS, Principal Investigator — Midwest Eye Center; J. Charles Henry, MD, Principal Investigator — Little Rock Eye Clinic; Elizabeth D. Sharpe, MD, Principal Investigator — Glaucoma Consultants & Center for Eye Research
Locations (5):
- United States (5):
  - Little Rock Eye Clinic, Little Rock, Arkansas
  - Omni Eye Services, Atlanta, Georgia
  - Midwest Eye Center, Bourbonnais, Illinois
  - Mark J. Weiss, MD, Tulsa, Oklahoma
  - Glaucoma Consultants & Center for Eye Research, Mt. Pleasant, South Carolina